CLINICAL TRIAL: NCT00735969
Title: High Dose Ribavirin in Combination With Peginterferon for Patients With Chronic Hepatitis C Genotype 1 Infection Who Have Failed to Respond or Relapsed After Standard Therapy
Brief Title: High-Dose Ribavirin and Peginterferon to Treat Chronic Hepatitis C Genotype 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marc Ghany, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080149; 08-DK-0149 (Other: NIH)
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2014-09-16 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Hepatitis C
Keywords: Non-Responder; Relapser; High Dose Ribavirin; Peginterferon; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Peginterferon
Drug: Ribavirin

SUMMARY:
This study will evaluate the effectiveness of an experimental treatment regimen for hepatitis C (HCV). Standard treatment consists of combination therapy with ribavirin, taken by mouth twice a day, and Peginterferon, injected under the skin once a week. Hepatitis C genotypes 2 and 3 have a high success rate with this regimen, while genotype 1 is more difficult to treat. This study will determine if patients with genotype 1 respond better to treatment that uses a higher dose of ribavirin than the standard approved dose of 1,000 to 1,200 mg daily.

Patients 18 years of age and older with chronic hepatitis C genotype 1 who have not been successfully treated with a standard course of Peginterferon and ribavirin may be eligible for this study. Participants eligible will receive Peginterferon plus twice the standard dose of ribavirin (2,000 to 2,400 mg daily) for 48 weeks. In addition to treatment, all patients receive undergo the following:

Before Treatment:

* Medical history and physical examination, symptom questionnaires, blood tests, urine collection, chest x-ray, electrocardiogram, liver ultrasound, Fibroscan (ultrasound to measure stiffness of the liver) and pregnancy test for women who are able to have children.
* Patients with other medical conditions or special risk factors may have further evaluations before starting treatment. These may include, for example, eye evaluation for patients with diabetes, exercise stress test for people over age 40 or who have risk factors for heart disease and psychiatric evaluation for people who have depression or anxiety disorder.

During Treatment

* Periodic blood tests to monitor blood counts and viral levels.
* Outpatient clinic visits every 4 weeks for the duration of the study for laboratory tests and review of symptoms and treatment side effects. Physical examinations and urine tests are done every 12 weeks.

Following Completion of Treatment

About 1 1/2 years after starting treatment, subjects are re-evaluated as they were at the start of treatment.

...

DETAILED DESCRIPTION:
Up to 60 patients with chronic hepatitis C genotype 1 infection who were previously treated with standard doses of peginterferon and ribavirin (1000 to 1200 mg daily) but who did not have a virological response (non-responders: n=35) or who relapsed after therapy (relapsers: n = 25) will be re-treated using peginterferon and higher doses of ribavirin (2000 to 2400 mg daily). After medical evaluation, documentation of eligibility and written informed consent, patients will be started on therapy with standard doses of peginterferon alfa-2a (180 micro g per week) and twice the standard dose of ribavirin (2000 mg daily for patients less than 75 kg; 2400 mg daily for patients greater than or equal to 75 kg). Viral kinetics will be evaluated on the basis of changes in HCV RNA levels during the first 24 weeks of therapy with blood sampling done on days 0, 1, and 2 and weeks 1, 2, 3, 4, 8, 12, 16, 20 and 24. Patients who fail to decrease levels of HCV RNA by more than 2 log(10) IU/ml by week 12 will be considered non-responders and therapy will stop. Similarly, patients who do not become HCV RNA negative (less than 10 IU) by week 24 will also be considered non-responders and therapy will be discontinued. Patients who do become HCV RNA negative during the first 24 weeks of therapy will continue for 48 weeks and be followed for at least 24 weeks thereafter. The primary end-point of this study will be a sustained virological response (SVR), which is defined by the absence of detectable HCV RNA in serum on treatment and for at least 24 weeks after stopping therapy. The SVR rate for re-treatment using conventional doses of peginterferon and ribavirin is expected to be less than 5 percent. The estimated rate of SVR using peginterferon with high doses of ribavirin is 50 percent for patients with a previous relapse and 25 percent for those with a previous non-response. A sample size of 35 patients would be needed to achieve statistical significance based upon these estimates of response rates for non-responders and 25 patients for relapsers. If none of the first ten non-responder patients treated in this protocol achieve an SVR, no more non-responder patients will be enrolled and this part of the study will be terminated early. Patients also will be monitored closely for side effects of therapy, the major one for ribavirin being anemia. Patients who develop anemia will be treated with darbepoietin to maintain a hemoglobin level above 10 gm percent. This pilot study is expected to demonstrate whether use of high doses of ribavirin is an option for patients who fail to have an adequate response to conventional doses of peginterferon and ribavirin for chronic hepatitis C.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18 years or above, male or female

Documented relapse or non-response to a prior adequate course of peginterferon and ribavirin

Genotype 1 HCV as determined by probe specific hybridization (Inno-Lipa assay).

Written informed consent.

EXCLUSION CRITERIA:

Age greater than 65 years

If cirrhosis is present, decompensated liver disease, as marked by serum bilirubin greater than 4 mg percent, albumin less than 3.0 gm percent, prothrombin time greater than 2 sec prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy.

Serum Alanine transaminase (ALT) or Aspartate transaminase (AST) levels greater than 1000 U/L (greater than 25 times the ULN). Such patients will not be enrolled but may be followed until three determinations are below this level.

Pregnancy or, in women of child bearing potential or in spouses of pregnant women, inability to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicide, or birth control pills, or an intrauterine device.

Breastfeeding.

Significant systemic or major illnesses including congestive heart failure, organ transplantation, serious psychiatric disease or depression, human immunodeficiency virus (HIV) infection, and angina pectoris.

Previous intolerance of weight based ribavirin dose (1,000-1,200 mg daily) including need for dose reduction, use of erythropoietin or serious adverse event attributable to ribavirin use.

Renal insufficiency (creatinine clearance less than 60 ml/min) or renal failure

Pre existing anemia (hematocrit less than 34 percent) or known history of hemolytic anemia.

Uncontrolled hypertension or diabetes mellitus

Other antiviral therapy within the last 6 months.

Immunosuppressive therapy with either corticosteroids (more than 5 mg of prednisone daily) or major immunosuppressive agents (such as azathioprine or 6-mercaptopurine).

Evidence of another form of liver disease in addition to viral hepatitis (for example autoimmune liver disease, Wilson disease, alcoholic liver disease, hemochromatosis, alpha 1 antitrypsin deficiency).

Evidence of coronary artery disease or cerebral vascular disease, including abnormalities on exercise stress testing in patients with defined risk factors who will be screened for evidence of underlying coronary artery disease.

Active substance abuse, such as alcohol, inhaled or injection drugs within the previous year.

Evidence of hepatocellular carcinoma; either alpha-fetoprotein (AFP) levels greater than 200 ng/ml (normal less than 9 ng/ml) and/or ultrasound (or other imaging study) demonstrating a mass suggestive of liver cancer.

Clinical gout.

Active, serious autoimmune disease, such as lupus erythematosis, ulcerative colitis, Crohn s disease or rheumatoid arthritis that in the opinion of the investigators might be exacerbated by therapy with peginterferon.

Uncontrolled thyroid disease

Evidence if severe retinopathy or clinically relevant ophthalmological disorder (only patients with pre-existing hypertension or diabetes will undergo an ophthalmological assessment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Liang TJ, Rehermann B, Seeff LB, Hoofnagle JH. Pathogenesis, natural history, treatment, and prevention of hepatitis C. Ann Intern Med. 2000 Feb 15;132(4):296-305. doi: 10.7326/0003-4819-132-4-200002150-00008. PMID 10681285
- [Background] Armstrong GL, Wasley A, Simard EP, McQuillan GM, Kuhnert WL, Alter MJ. The prevalence of hepatitis C virus infection in the United States, 1999 through 2002. Ann Intern Med. 2006 May 16;144(10):705-14. doi: 10.7326/0003-4819-144-10-200605160-00004. PMID 16702586
- [Background] Nainan OV, Alter MJ, Kruszon-Moran D, Gao FX, Xia G, McQuillan G, Margolis HS. Hepatitis C virus genotypes and viral concentrations in participants of a general population survey in the United States. Gastroenterology. 2006 Aug;131(2):478-84. doi: 10.1053/j.gastro.2006.06.007. PMID 16890602
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-DK-0149.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginterferon and Ribavirin Arm: Patients 18 years of age and older with chronic hepatitis C genotype 1 who have not been successfully treated with a standard course of Peginterferon and ribavirin are screened and assigned to receive Peginterferon plus twice the dose of ribavirin (2,000 to 2,400 mg daily) for 48 weeks.
Period: Overall Study
Arm/Group | Peginterferon and Ribavirin Arm
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients 18 years of age and older with chronic hepatitis C genotype 1 who have not been successfully treated with a standard course of Peginterferon and ribavirin.
Groups:
- Peginterferon and Ribavirin Arm: Patients 18 years of age and older with chronic hepatitis C genotype 1 who have not been successfully treated with a standard course of Peginterferon and ribavirin are screened and randomly assigned to receive either standard treatment with Peginterferon and ribavirin or to receive Peginterferon plus twice the dose of ribavirin (2,000 to 2,400 mg daily) for 48 weeks.
Arm/Group | Peginterferon and Ribavirin Arm
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response, (HCV RNA Neg.) in Serum 24 Weeks Off Therapy.
Time Frame: 24 weeks after treatment stop
Measure: Number; unit: participants
Arm/Group | Peginterferon and Ribavirin Arm
Number analyzed (Participants) | 21
participants | 3

ADVERSE EVENTS:
Arm/Group | Peginterferon and Ribavirin Arm
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon and Ribavirin Arm (N=21)
symptomatic anemia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes